CLINICAL TRIAL: NCT01865747
Title: A Phase 3, Randomized, Controlled Study of Cabozantinib (XL184) vs Everolimus in Subjects With Metastatic Renal Cell Carcinoma That Has Progressed After Prior VEGFR Tyrosine Kinase Inhibitor Therapy
Brief Title: A Study of Cabozantinib (XL184) vs Everolimus in Subjects With Metastatic Renal Cell Carcinoma
Acronym: METEOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-308
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell cancer; kidney; vascular endothelial growth factor receptor 2 (VEGFR2); tyrosine kinase inhibitor; hepatocyte growth factor receptor protein (MET); von Hippel-Lindau gene
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Everolimus; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib (XL184) (Experimental): Cabozantinib (XL184) 60 mg tablet once daily.
  Interventions: Drug: Cabozantinib tablets
- Everolimus (Afinitor) (Active Comparator): Everolimus (Afinitor) 10 mg tablet once daily.
  Interventions: Drug: Everolimus (Afinitor) tablets

INTERVENTIONS:
Drug: Cabozantinib tablets
  Other Names: XL184
  Arms: Cabozantinib (XL184)
Drug: Everolimus (Afinitor) tablets
  Arms: Everolimus (Afinitor)

SUMMARY:
The purpose of this study is to evaluate the effect of Cabozantinib (XL184) compared with Everolimus (Afinitor) on progression-free survival (PFS) and overall survival (OS) in subjects with advanced renal cell cancer that has progressed after prior VEGFR tyrosine kinase inhibitor therapy.

ELIGIBILITY:
Select Inclusion Criteria:

1. Documented histological or cytological diagnosis of renal cell cancer with a clear-cell component.
2. Measurable disease as determined by the investigator.
3. Must have received at least one VEGFR-targeting TKI (eg, sorafenib, sunitinib, axitinib, pazopanib or tivozanib).
4. Recovery from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
5. Adequate organ and marrow function.
6. Sexually active fertile subjects(male and female)must agree to use medically accepted methods of contraception during the course of the study and for 4 months after the last dose of study treatment.
7. Female subjects of childbearing potential must not be pregnant at screening.

Select Exclusion Criteria:

1. Prior treatment with everolimus, or any other specific or selective TORC1/PI3K/AKT inhibitor (eg, temsirolimus), or cabozantinib.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before randomization.
3. Receipt of any type of anticancer antibody (including investigational antibody) within 4 weeks before randomization.
4. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before randomization. Systemic treatment with radionuclides within 6 weeks before randomization. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before randomization.
6. Concomitant anticoagulation at therapeutic doses with oral anticoagulants or platelet inhibitors.
7. Chronic treatment with corticosteroids or other immunosuppressive agents.
8. Serious illness other than cancer.
9. Major surgery within 3 months before randomization. Complete wound healing from major surgery must have occurred 1 month before randomization and from minor surgery at least 10 days before randomization.
10. Pregnant or lactating females.
11. Diagnosis of another malignancy within 2 years before randomization, except for superficial skin cancers, or localized, low grade tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05-22 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (184):
- United States (49):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Vallejo, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Westwood, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Albany, New York
  - New York, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Vancouver, Washington
  - Yakima, Washington
- Argentina (2):
  - La Plata, Buenos Aires
  - Mar del Plata
- Australia (14):
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Kogarah, New South Wales
  - Port Macquarie, New South Wales
  - Randwick, New South Wales
  - Wahroonga, New South Wales
  - Westmead, New South Wales
  - Milton, Queensland
  - Wooloongabba, Queensland
  - Adelaide, South Australia
  - Hobart, Tasmania
  - Bentleight East, Victoria
  - Box Hill, Victoria
  - Wodonga, Victoria
- Austria (2):
  - Linz, Upper Austria
  - Vienna
- Belgium (7):
  - Bonheiden, Antwerpen
  - Brasschaat, Antwerpen
  - Brussels, Brussels Capital
  - Leuven, Vlaams Brabant
  - Roeselare, West-Vlaanderen
  - Antwerp
  - Liège
- Canada (13):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnepeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Santiago, Chile
- Czechia (3):
  - Olomouc, Olomoucký kraj
  - Brno
  - Prague
- Denmark (3):
  - Herlev, Capital Region
  - Aarhus, Central Jutland
  - Odense, Region Syddanmark
- Finland (2):
  - Turku, Länsi-Suomen Lääni
  - Helsinki
- France (11):
  - Caen, Calvados
  - Besançon, Doubs
  - Bordeaux, Gironde
  - Toulouse, Haute-Garonne
  - Rennes, Ille-et-Vilaine
  - Nantes, Loire-Atlantique
  - Lyon, Rhône
  - Le Mans, Sarthe
  - Villejuif, Val-de-Marne
  - Marseille
  - Paris
- Germany (18):
  - Freiburg im Breisgau, Baden Wuttemberg
  - Tübingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Aachen, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Erfurt, Thuringia
  - Jena, Thuringia
  - Berlin
  - Dresden
  - Frankfurt am Main
  - Gütersloh
  - Hamburg
  - Hanover
  - Heidelberg
  - Munich
  - München
- Hungary (2):
  - Budapest
  - Szolnok
- Dublin, Ireland
- Italy (9):
  - Bari, Apulia
  - Meldola, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Ravenna, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Cremona, Lombardy
  - Arezzo, Tuscany
  - Terni, Umbria
- Netherlands (4):
  - Maastricht, Limburg
  - Amsterdam, North Holland
  - Leiden, South Holland
  - Rotterdam, South Holland
- Poland (4):
  - Poznan, Greater Poland Voivodeship
  - Bialystok, Podlaskie Voivodeship
  - Gdansk, Pomeranian Voivodeship
  - Warsaw
- Portugal (2):
  - Lisbon
  - Porto
- Russia (4):
  - Moscow
  - Omsk
  - Saint Petersburg
  - Yaroslavl
- Slovakia (2):
  - Prešov
  - Žilina
- Seoul, South Korea
- Spain (11):
  - Badalona, Catalonia
  - Barcelona, Catalonia
  - L'Hospitalet de Llobregat, Catalonia
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Barcelona
  - Madrid
  - Málaga
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (3):
  - Lund, Skåne County
  - Stockholm, Södermanland County
  - Umeå
- Taiwan (2):
  - Taichung
  - Taipei
- Turkey (Türkiye) (4):
  - Ankara
  - Gaziantep
  - Istanbul
  - Izmir
- United Kingdom (10):
  - Birmingham, England
  - Derby, England
  - Guildford, England
  - London, England
  - Manchester, England
  - Metropolitan Borough of Wirral, England
  - Northwood, England
  - Aberdeen, Scotland
  - Edinburgh, Scotland
  - Glasgow, Scotland

REFERENCES:
- [Derived] Gong AJ, Ruchalski K, Kim HJ, Douek M, Gutierrez A, Patel M, Sai V, Coy H, Villegas B, Raman S, Goldin J. RECIST 1.1 Target Lesion Categorical Response in Metastatic Renal Cell Carcinoma: A Comparison of Conventional versus Volumetric Assessment. Radiol Imaging Cancer. 2023 Sep;5(5):e220166. doi: 10.1148/rycan.220166. PMID 37656041
- [Derived] Denize T, Farah S, Cimadamore A, Flaifel A, Walton E, Sticco-Ivins MA, Labaki C, Braun DA, Sun M, Wang E, Xie W, Choueiri TK, Signoretti S. Biomarkers of Angiogenesis and Clinical Outcomes to Cabozantinib and Everolimus in Patients with Metastatic Renal Cell Carcinoma from the Phase III METEOR Trial. Clin Cancer Res. 2022 Feb 15;28(4):748-755. doi: 10.1158/1078-0432.CCR-21-3088. PMID 34921022
- [Derived] Powles T, Choueiri TK, Motzer RJ, Jonasch E, Pal S, Tannir NM, Signoretti S, Kaldate R, Scheffold C, Wang E, Aftab DT, Escudier B, George DJ. Outcomes based on plasma biomarkers in METEOR, a randomized phase 3 trial of cabozantinib vs everolimus in advanced renal cell carcinoma. BMC Cancer. 2021 Aug 7;21(1):904. doi: 10.1186/s12885-021-08630-w. PMID 34364385
- [Derived] Donskov F, Motzer RJ, Voog E, Hovey E, Grullich C, Nott LM, Cuff K, Gil T, Jensen NV, Chevreau C, Negrier S, Depenbusch R, Bergmann L, Cornelio I, Champsaur A, Escudier B, Pal S, Powles T, Choueiri TK. Outcomes based on age in the phase III METEOR trial of cabozantinib versus everolimus in patients with advanced renal cell carcinoma. Eur J Cancer. 2020 Feb;126:1-10. doi: 10.1016/j.ejca.2019.10.032. Epub 2019 Dec 27. PMID 31887537
- [Derived] Flaifel A, Xie W, Braun DA, Ficial M, Bakouny Z, Nassar AH, Jennings RB, Escudier B, George DJ, Motzer RJ, Morris MJ, Powles T, Wang E, Huang Y, Freeman GJ, Choueiri TK, Signoretti S. PD-L1 Expression and Clinical Outcomes to Cabozantinib, Everolimus, and Sunitinib in Patients with Metastatic Renal Cell Carcinoma: Analysis of the Randomized Clinical Trials METEOR and CABOSUN. Clin Cancer Res. 2019 Oct 15;25(20):6080-6088. doi: 10.1158/1078-0432.CCR-19-1135. Epub 2019 Aug 1. PMID 31371341
- [Derived] Cella D, Escudier B, Tannir NM, Powles T, Donskov F, Peltola K, Schmidinger M, Heng DYC, Mainwaring PN, Hammers HJ, Lee JL, Roth BJ, Marteau F, Williams P, Baer J, Mangeshkar M, Scheffold C, Hutson TE, Pal S, Motzer RJ, Choueiri TK. Quality of Life Outcomes for Cabozantinib Versus Everolimus in Patients With Metastatic Renal Cell Carcinoma: METEOR Phase III Randomized Trial. J Clin Oncol. 2018 Mar 10;36(8):757-764. doi: 10.1200/JCO.2017.75.2170. Epub 2018 Jan 29. PMID 29377755
- [Derived] Escudier B, Powles T, Motzer RJ, Olencki T, Aren Frontera O, Oudard S, Rolland F, Tomczak P, Castellano D, Appleman LJ, Drabkin H, Vaena D, Milwee S, Youkstetter J, Lougheed JC, Bracarda S, Choueiri TK. Cabozantinib, a New Standard of Care for Patients With Advanced Renal Cell Carcinoma and Bone Metastases? Subgroup Analysis of the METEOR Trial. J Clin Oncol. 2018 Mar 10;36(8):765-772. doi: 10.1200/JCO.2017.74.7352. Epub 2018 Jan 8. PMID 29309249
- [Derived] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Derived] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 08 August 2013, Data cut off date: 22 May 2015
Groups:
- Cabozantinib (XL184): Cabozantinib (XL184) 60 mg tablet once daily.
  Cabozantinib tablets
- Everolimus (Afinitor): Everolimus (Afinitor) 10 mg tablet once daily.
  Everolimus (Afinitor) tablets
Period: Overall Study (ITT)
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Started (Randomized) | 330 | 328
Completed (Continuing study treatment at the time of data cut-off) | 132 (One subject randomized to everolimus arm received cabozantinib discontd due to clin. deterioration) | 73 (Five subjects were randomized but not treated)
Not Completed | 198 | 255
Not completed — Adverse Event | 32 | 31
Not completed — Clinical Deterioration | 29 | 50
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Sponsor Decision | 0 | 1
Not completed — Progressive Disease | 122 | 158
Not completed — Reason Not Provided | 0 | 1
Period: Primary Intent to Treat (PITT)
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Started (PITT population consisted of the first 375 subjects randomized to received study treatment.) | 187 | 188 (Three subjects in the everolimus arm were randomized but not treated.)
Completed (Continuing study treatment at the time of data cut-off) | 56 | 36
Not Completed | 131 | 152
Not completed — Adverse Event | 21 | 20
Not completed — Clinical Deterioration | 18 | 29
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Progressive Disease | 82 | 92
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor) | Total
Number analyzed (Participants) | 330 | 328 | 658
Age, Customized [Number; unit: participants]
  <65 | 196 | 198 | 394
  65 to <75 | 107 | 94 | 201
  75 to <85 | 26 | 36 | 62
  =>85 | 1 | 0 | 1
Sex/Gender, Customized [Number; unit: participants]
  Male | 253 | 241 | 494
  Female | 77 | 86 | 163
  Missing | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 19 | 18 | 37
  Ethnicity: Not Hispanic or Latino | 278 | 273 | 551
  Ethnicity: Unknown or Not Reported | 33 | 37 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 26 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 269 | 263 | 532
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 34 | 36 | 70
Geographic Region [Count of Participants; unit: Participants]
  Europe | 167 | 153 | 320
  North America | 118 | 122 | 240
  Asia Pacific | 39 | 47 | 86
  Latin America | 6 | 6 | 12
Randomization Stratification Factors per CRF [Count of Participants; unit: Participants]
  Prior VEGFR-TKI = 1 | 235 | 229 | 464
  Prior VEGFR-TKI ≥ 2 | 95 | 99 | 194
  MSKCC risk factors = 0 | 150 | 150 | 300
  MSKCC risk factors = 1 | 139 | 135 | 274
  MSKCC risk factors = 2 or 3 | 41 | 43 | 84
  Prior VEGFR-TKI = 1, MSKCC risk factors = 0 | 102 | 100 | 202
  Prior VEGFR-TKI = 1, MSKCC risk factors = 1 | 107 | 103 | 210
  Prior VEGFR-TKI = 1, MSKCC risk factors = 2 or 3 | 26 | 26 | 52
  Prior VEGFR-TKI ≥ 2, MSKCC risk factors =0 | 48 | 50 | 98
  Prior VEGFR-TKI ≥ 2, MSKCC risk factors = 1 | 32 | 32 | 64
  Prior VEGFR-TKI ≥ 2, MSKCC risk factors = 2 or 3 | 15 | 17 | 32
Karnofsky performance status (KPS) [Count of Participants; unit: Participants]
  100 (normal activity) | 99 | 74 | 173
  90 (normal activity, minor signs and symptoms) | 127 | 142 | 269
  80 (normal w/effort, minor signs/symptoms) | 75 | 90 | 165
  70 (unable to work, cares for self) | 29 | 22 | 51
Heng Prognostic Criteria [Count of Participants; unit: Participants]
  0 adverse factors (favorable risk) | 66 | 62 | 128
  1-2 adverse factors (intermediate risk) | 210 | 214 | 424
  3-6 adverse factors (poor risk) | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The primary analysis of PFS is the time from randomization to date of first documented tumor progression as determined by investigator (per RECIST 1.1 criteria) or death due to any cause, whichever occurred first. A Kaplan-Meier analysis was performed to estimate the median duration.
Time Frame: PFS is measured from the date of randomization until the date of first documented disease progression or date of death from any cause as determined by the Independent Radiology Committee (IRC) per RECIST 1.1, assessed for up to 17 months.
Population: The pre-specified primary analysis of PFS was based on the first 375 randomized subjects (187 cabozantinib and 188 everolimus).
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Number analyzed (Participants) | 187 | 188
months | 7.4 [5.6 to 9.1] | 3.8 [3.7 to 5.4]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Everolimus (Afinitor); Test type: Superiority; p < 0.0001, Log Rank; The Log-Rank Test was stratified by the Memorial Sloan-Kettering Cancer Center (MSKCC) group and number of prior VEGFR TKIs; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.45 to 0.74]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from randomization to the date of death. Participants that had not died were censored at last known date alive. Median OS was calculated using Kaplan-Meier estimates. Interim analyses for OS occurred after 320 deaths (78% of the total OS events needed for final analysis).
Time Frame: OS was measured from the time of randomization until 320 deaths, approximately 28 months
Population: The Intent to Treat (ITT) population was used and included 658 randomized subjects (330 cabozantinib, 328 everolimus) in the second interim analysis with a cutoff date of 31 December 2015.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Number analyzed (Participants) | 330 | 228
months | 21.4 [18.7 to NA] — Too few events to estimate the upper limit of the confidence interval. | 16.5 [14.7 to 18.8]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Everolimus (Afinitor); Test type: Superiority; p = 0.0003, Log Rank; The Log-Rank test was stratified by the Memorial Sloan-Kettering Cancer Center (MSKCC) risk group and number of prior VEGFR TKIs; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.53 to 0.83]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is the number of participants with a best response of complete response (CR) or partial response (PR) divided by number of randomized participants. ORR was assessed by the Independent Radiology Committee (IRC) per RECIST 1.1 which was confirmed by a subsequent visit >= 28 days later, and was analyzed in the Intent to Treat (ITT) population at the time of the primary analysis of Progression Free Survival (PFS). The data cutoff date was 22 May 2015.
Time Frame: ORR was assessed at 8 weeks post-randomization, every 8 weeks for 12 months, and every 12 weeks until date of disease progression or death, up to May 2015 (approximately 21 months)
Population: The analysis of ORR was performed in the ITT population (all randomized: 330 cabozantinib, 328 everolimus) based upon response determined by Independent Radiology Committee (IRC) per RECIST 1.1.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Number analyzed (Participants) | 330 | 328
percentage of participants | 17 | 3
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Everolimus (Afinitor); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 08 August 2013 - 22 May 2015
Description: The safety data includes subjects who were randomized and treated. Of 658 patients, 330 were randomized to receive cabozantinib and 328 everolimus. Five subjects in the everolimus arm were randomized but not treated. One subject randomized to the everolimus arm received cabozantinib only as study treatment and was evaluated in the cabozantinib arm for the Safety population (331 cabozantinib, 322 everolimus).
Arm/Group | Cabozantinib (XL184) | Everolimus (Afinitor)
Serious Adverse Events (participants affected / at risk) | 131/331 | 139/322
Other Adverse Events (participants affected / at risk) | 328/331 | 270/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (XL184) (N=331) | Everolimus (Afinitor) (N=322)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 12 (12)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypercalcaemia of Malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 10 (10) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Oesophageal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestine Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Asthenia (General disorders) | 4 (4) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Device Occlusion (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 5 (5)
General Physical Health Deterioration (General disorders) | 4 (4) | 6 (6)
Generalised Oedema (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 2 (2)
Mutli-Organ Failure (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Ulcer Haemorrhage (General disorders) | 1 (1) | 0 (0)
Bile Duct Obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis Cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess Neck (Infections and infestations) | 0 (0) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 2 (2) | 0 (0)
Anorectal Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 1 (1) | 0 (0)
Aspergillus Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pleural Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 13 (13)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Vulval Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foreign Body in Eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Blood Cholesterol Increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm of Orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Metastases to Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metatases to Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metatases to Testicle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 11 (11)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour Thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Venous Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Miller Fisher Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 1 (1) | 4 (4)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 5 (5)
Renal Haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (XL184) (N=331) | Everolimus (Afinitor) (N=322)
Hypothyroidism (Endocrine disorders) | 68 (68) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 50 (50) | 30 (30)
Abdominal Pain Upper (Gastrointestinal disorders) | 26 (26) | 7 (7)
Constipation (Gastrointestinal disorders) | 83 (83) | 61 (61)
Diarrhoea (Gastrointestinal disorders) | 245 (245) | 88 (88)
Dyspepsia (Gastrointestinal disorders) | 40 (40) | 15 (15)
Flatulence (Gastrointestinal disorders) | 32 (32) | 6 (6)
Nausea (Gastrointestinal disorders) | 164 (164) | 89 (89)
Vomiting (Gastrointestinal disorders) | 105 (105) | 44 (44)
Fatigue (General disorders) | 185 (185) | 149 (149)
Alanine Aminotransferase Increased (Investigations) | 53 (53) | 19 (19)
Aspartate Aminotransferase Increased (Investigations) | 58 (58) | 18 (18)
Blood Thyrpod Stimulating Hormone Increased (Investigations) | 23 (23) | 3 (3)
Weight Decreased (Investigations) | 104 (104) | 39 (39)
Decreased Appetite (Metabolism and nutrition disorders) | 152 (152) | 108 (108)
Hypomagnesaemia (Metabolism and nutrition disorders) | 50 (50) | 5 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 42 (42) | 16 (16)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 46 (46) | 25 (25)
Dysgeusia (Nervous system disorders) | 78 (78) | 30 (30)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 66 (66) | 12 (12)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 139 (139) | 19 (19)
Hypertension (Vascular disorders) | 122 (122) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.